CLINICAL TRIAL: NCT04304820
Title: Early Initiation of Oral Therapy With Cyclosporine and Eltrombopag for Treatment Naive Severe Aplastic Anemia (SAA)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200033; 20-H-0033
Record Dates: First submitted 2020-03-10; First posted 2020-03-11 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Severe Aplastic Anemia
Keywords: Immunosuppression; T-cells; Hematopoiesis; Autoimmunity; Thrombocytopenia
MeSH Terms: conditions — Anemia, Aplastic; Autoimmune Diseases; Thrombocytopenia | interventions — eltrombopag; Cyclosporine; Antilymphocyte Serum

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with Severe Aplastic Anemia in Early Initiation of Cyclosporine and Eltrombopag (Experimental): Treatment-naïve Severe Aplastic Anemia (SAA) participants start Cyclosporine (CsA) on Day 1 at 2 mg/kg/day. At initiation of Horse Anti-Thymocyte-Globulin (h-ATG), dosing increases to 3 mg/kg every 12 hours for those ≥12 years (6 mg/kg/day total) and 6 mg/kg every 12 hours for those <12 years (12 mg/kg/day total). Actual body weight is used unless >125% ideal body weight (IBW), where adjusted IBW applies. CsA is titrated to a trough of 200-400 mcg/L. At 6 months, responders reduce to 2 mg/kg/day through 24 months, with return to full dosing if relapse occurs. h-ATG is given at 40 mg/kg/day for 4 days IV, unless the patient already shows a complete response at the initial NIH visit after remote oral therapy.
  Eltrombopag (EPAG) starts on Day 1 at 150 mg/day for ages 12-17, 75 mg/day for ages 6-11, and 2.5 mg/kg/day for ages 3-5. For East and Southeast Asian patients, starting doses are reduced to 75 mg/day (ages 12-85), 37.5 mg/day (ages 6-11), and 1.25 mg/kg/day (ages 3-5).
  Interventions: Drug: Eltrombopag; Drug: Cyclosporine; Drug: Horse-Anti-thymocyte-Globulin
- Extension Cohort (Experimental): Treatment-naïve Severe Aplastic Anemia (SAA) participants start Cyclosporine (CsA) on Day 1 at 2 mg/kg/day. At initiation of Horse Anti-Thymocyte-Globulin (h-ATG), dosing increases to 3 mg/kg every 12 hours for those ≥12 years (6 mg/kg/day total) and 6 mg/kg every 12 hours for those <12 years (12 mg/kg/day total). Actual body weight is used unless >125% ideal body weight (IBW), where adjusted IBW applies. CsA is titrated to a trough of 200-400 mcg/L. At 6 months, responders reduce to 2 mg/kg/day through 24 months, with return to full dosing if relapse occurs. h-ATG is given at 40 mg/kg/day for 4 days IV, unless the patient already shows a complete response at the initial NIH visit after remote oral therapy.
  Eltrombopag (EPAG) starts on Day 1 at 150 mg/day for ages 12-17, 75 mg/day for ages 6-11, and 2.5 mg/kg/day for ages 3-5. For East and Southeast Asian patients, starting doses are reduced to 75 mg/day (ages 12-85), 37.5 mg/day (ages 6-11), and 1.25 mg/kg/day (ages 3-5).
  Interventions: Drug: Eltrombopag; Drug: Cyclosporine; Drug: Horse-Anti-thymocyte-Globulin

INTERVENTIONS:
Drug: Eltrombopag — Between 12 and 17yo (adult dose of 150mg) Between 6 and 11yo (75 mg) Between 3 and 5 yo (2.5 mg/kg)
  Other Names: EPAG
Drug: Cyclosporine — Day 1 to start of h-ATG: 2mg/kg/day by mouth (All subjects) Start of h-ATG to Month 6: 3 mg/kg/dose by mouth administered every 12 hours (12yo and above) 6 mg/kg/dose by mouth administered every 12 hours (less than 12yo) Month 6 to Month 24: Dosing to be adjusted based on response
  Other Names: CsA
Drug: Horse-Anti-thymocyte-Globulin — h-ATG at a dose of 40 mg/kg/day for 4 days (intravenously for approximately 4 hours daily) Note: Omitted in patients who have achieved a complete response at the initial NIH visit after initiating oral treatment remotely
  Other Names: H-ATG

SUMMARY:
Background:

Severe aplastic anemia (SAA) is a rare and serious blood disorder. It causes the immune system to turn against bone marrow cells. Standard treatment for SSA is a combination of 3 drugs (Cyclosporine [CsA], Eltrombopag [EPAG], and horse anti-thymocyte globulin [h-ATG]). Researchers want to see if starting people at a lower dose of CsA with EPAG before giving them h-ATG is helpful.

Objective:

To learn if early initiation of oral therapy with CsA and EPAG is safe and effective in people who have SAA and have not been treated with a course of immunosuppressive therapy and EPAG.

Eligibility:

People ages 3 and older with SAA

Design:

Participants will be screened with:

* medical history
* physical exam
* electrocardiogram
* blood tests
* family history
* bone marrow biopsy
* current medicines.

Participants may be screened remotely via telephone conference.

Participants will take a lower oral dose of CsA and EPAG. They will take CsA twice a day for 6 months. They will take EPAG for 6 months. Those who cannot visit the NIH Clinical Center within 72 hours will start taking the drugs at home. They will have weekly telephone calls with NIH staff until they visit the Clinical Center.

Participants may get h-ATG at the Clinical Center for 4 days. For this, they will have a central line placed. It is a plastic tube inserted into a neck, chest, or arm vein.

Participants will repeat most screening tests throughout the study.

Participants will have follow-up visits at the Clinical Center at 3 months, 6 months, and annually for 5 years after the start of the study....

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a life-threatening bone marrow failure characterized by pancytopenia and a hypocellular marrow. Allogeneic bone marrow transplantation is curative in younger patients, but older age and/or lack of a suitable donor have limited application of this procedure. As an alternative to transplant, immunosuppressive treatment (IST) has provided durable remissions and similar long term survival [1]. Approximately 2/3 of patients who receive IST with horse anti-thymocyte globulin (h-ATG) and cyclosporine (CsA) have blood count recovery, but 25-30% do not respond and 30-40% will relapse. A likely explanation for partial recovery and relapse is incomplete elimination of auto-reactive T cells and insufficient stem cell reserve.

Thrombopoietin (TPO) is a key regulator of hematopoietic stem cell renewal and survival. To improve the hematologic response rate, our group assessed the addition of eltrombopag (EPAG), a synthetic mimetic of TPO, to IST in treatment na(SqrRoot) ve SAA. This combination achieved a higher complete response rate to about 50% and an overall response rate to 80%, both superior to historic controls [2]. This regimen received FDA approval in November 2018. Combined therapy is now being tested in a European randomized study. Furthermore, protocols have been developed internationally to determine whether EPAG and CsA, without ATG, are sufficient to improve blood counts, in countries where ATG is not available.

The long-term complications, relapse and clonal evolution, were no worse with the addition of EPAG than in our historical cohort, but still remain a problem. Clonal evolution occurs in 10-15% of patients and is defined as development of myelodysplastic syndrome or acute myeloid leukemia with characteristic cytogenetic abnormalities of aneuploidy, especially monosomy 7 or deletion 7q. There are no predictive tools to identify patients at higher risk for either of these two long term events.

Because SAA is a rare disease, treatment has been recommended to take place at a specialized center. However, delays in reaching such centers and initiating therapy are common. From current understanding of the disease, immune destruction of cells is ongoing during this period, likely impacting on both short and long term outcomes. We propose early initiation of lower dose CsA (2mg/kg/day) and EPAG to decrease ongoing immune destruction and stimulate HSPC while awaiting full work up and transfer to the Clinical Center (CC).

The aim of this study is to test feasibility and safety of initiating oral therapy before arriving to the NIH, based on diagnostic tests performed by local physicians and interpretation from experts here. Treatment will be initiated remotely but under complete guidance and supervision of the research team at the Hematology Branch. All patients except the ones who achieve complete response will receive standard three drug regimen upon completion of work up here at the CC. Primary endpoint of the study will be to assess feasibility and safety as a composite measure of misdiagnosis, non-compliance with the regimen or failure to establish care at the Clinical Center within 8 weeks of initiating treatment, and TRSAE (treatment related serious adverse events). Initial treatment period of 8 weeks may be extended in special circumstances. Secondary endpoints are response rates at landmark time points, relapse, overall survival, and clonal evolution.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age >= 3 years old
  2. Weight >12Kg
  3. Severe aplastic anemia:
* Bone marrow cellularity <30% (excluding lymphocytes) AND At least two of the following:

  * Absolute neutrophil count <500/microliter
  * Platelet count <20,000/microliter
  * Absolute reticulocyte count <60,000/microliter

EXCLUSION CRITERIA:

1. Known diagnosis or high suspicion of Fanconi anemia or other constitutional marrow failure syndrome
2. Evidence of a clonal disorder on cytogenetics performed within 12 weeks of study entry involving chromosome 7 or complex karyotype. Patient will not be excluded if cytogenetics are not done or are pending
3. A course of prior immunosuppressive therapy (ATG, cyclosporine, alemtuzumab, and high dose cyclophosphamide), or eltrombopag
4. SGOT or SGPT >2.5 times the upper limit of normal or total bilirubin >1.5 x upper limit of normal
5. Subjects with liver cirrhosis (as determined by the investigator).
6. Subjects with human immunodeficiency virus (HIV) who are not receiving antiretroviral therapy, have detectable HIV RNA viral load and have CD4 cell count <200/microliter, or are on anti-retroviral therapy that interacts with the study drugs. subjects will not be excluded if HIV testing is pending or unavailable.
7. Glomerular filtration rate (GFR) <40 mL/min/1.73m^2
8. Hypersensitivity to EPAG or its components
9. Infection not adequately responding to appropriate therapy
10. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy, or that death within 7-10 days is likely
11. Potential subjects with cancer who are on active chemotherapeutic treatment or who take drugs with hematological effects will not be eligible
12. Inability to understand the investigational nature of the study or to give informed consent or does not have a legally authorized representative or surrogate that can provide informed consent.
13. Inability to swallow
14. Unable to participate in audio/video telecommunication
15. Inability to ship the study drug to participant
16. History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following: Recent myocardial infarction (within last 6 months), uncontrolled congestive heart failure, unstable angina (within last 6 months), clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker.), long QT syndrome, family history of idiopathic sudden death, congenital long QT syndrome or additional risk factors for cardiac repolarization abnormality, as determined by the investigator.
17. Impaired cardiac function, such as: Corrected QTc >450 msec using Fridericia correction (QTcF) on the screening ECG (using triplicate ECGs), other clinically significant cardiovascular disease (e.g., uncontrolled hypertension, history of labile hypertension), history of known structural abnormalities (e.g. cardiomyopathy).
18. Concurrent participation in an investigational study within 30 days prior to enrollment or within 5-half-lives of the investigational product, whichever is longer. Note: parallel enrollment in a disease registry is permitted.
19. Known thrombophilic risk factors. Exception: Subjects for whom the potential benefits of participating in the study outweigh the potential risks of thromboembolic events, as determined by the investigator.
20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of study treatment. Basic contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject
    * Barrier methods of contraception: Condom or Occlusive cap. For the UK: with spermicidal foam/gel/film/cream/ vaginal suppository
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

      * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
21. Female subjects who are nursing or pregnant (positive serum or urine B-human chorionic gonadotrophin (B-hCG) pregnancy test) at screening or pre-dose on Day 1
22. Sexually active males unless they use a condom during intercourse while taking the drug during treatment, and for 7 days after stopping treatment (and for an additional 12 weeks [for genotoxic compounds]) and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via semen.

INCLUSION OF PREGNANT WOMEN, FETUSES OR NEONATES:

The protocol does not intentionally enroll pregnant women due to unknown fetal risk with eltrombopag. However, if a patient gets pregnant during the trial participation period, she may remain on study for non-invasive safety and outcomes follow-up.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2033-12-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavisha A Patel, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting approximately 6 months after publication and available indefinitely.
Access Criteria: Data may be shared through an open or closed repository as appropriate.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-H-0033.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Severe Aplastic Anemia in Early Initiation of Cyclosporine and Eltrombopag: Treatment-naïve Severe Aplastic Anemia (SAA) participants start Cyclosporine (CsA) on Day 1 at 2 mg/kg/day. At initiation of Horse Anti-Thymocyte-Globulin (h-ATG), dosing increases to 3 mg/kg every 12 hours for those ≥12 years (6 mg/kg/day total) and 6 mg/kg every 12 hours for those <12 years (12 mg/kg/day total). Actual body weight is used unless >125% ideal body weight (IBW), where adjusted IBW applies. CsA is titrated to a trough of 200-400 mcg/L. At 6 months, responders reduce to 2 mg/kg/day through 24 months, with return to full dosing if relapse occurs. h-ATG is given at 40 mg/kg/day for 4 days IV, unless the patient already shows a complete response at the initial NIH visit after remote oral therapy.
  Eltrombopag (EPAG) starts on Day at 150 mg/day for ages 12-17, 75 mg/day for ages 6-11, and 2.5 mg/kg/day for ages 3-5. For East and Southeast Asian patients, starting doses are reduced to 75 mg/day (ages 12-85), 37.5 mg/day (ages 6-11), and 1.25 mg/kg/day (ages 3-5).
Period: Overall Study
Arm/Group | Participants With Severe Aplastic Anemia in Early Initiation of Cyclosporine and Eltrombopag
Started | 39
Completed | 28
Not Completed | 11
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Pursuing Stem Cell Transplant | 4
Not completed — Pursuing Additional Immunosuppressive therapy | 4
Not completed — Evolution to Myeloid Malignancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Severe Aplastic Anemia in Early Initiation of Cyclosporine and Eltrombopag
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 31
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 17
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting Safety and Feasibility Criteria During Study Treatment Period With Oral Treatment (Low Dose Cyclosporine and Eltrombopag) Until the Start of Standard of Care Treatment (Horse Anti-thymocyte-globulin)
Description: For the primary endpoint of this study, the treatment is defined to be "feasible" to a participant if he/she meets the safety and feasibility criteria. Safety and feasibility criteria is a composite measure of as defined as TRSAE, mis- and altered diagnosis, and non-compliance with the regimen or failure to establish care at the National Institutes of Health Clinical Center. Study treatment period is defined as the duration from the initiation of oral treatment (low dose Cyclosporine and Eltrombopag) to the start of standard of care treatment (horse anti-thymocyte-globulin).
Time Frame: Up to 12 Weeks from the initiation of oral treatment (Low Dose Cyclosporine and Eltrombopag)
Population: analysis was intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Severe Aplastic Anemia in Early Initiation of Cyclosporine and Eltrombopag
Number analyzed (Participants) | 39
Participants | 37

2. Secondary Outcome: Hematological Response
Time Frame: At 1, 2, 3, 6 and 12 months and yearly thereafter
Reporting Status: Not Posted

3. Secondary Outcome: Relapse
Time Frame: At 1, 2, 3, 6 and 12 months and yearly thereafter
Reporting Status: Not Posted

4. Secondary Outcome: Clonal Evolution to PNH, Clonal Chromosomal Population in Bone Marrow, Myelodysplasia by Morphology, or Acute Leukemia
Time Frame: At 1, 2, 3, 6 and 12 months and yearly thereafter
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Time Frame: At 5 Years (60 Months)
Reporting Status: Not Posted

6. Secondary Outcome: Hematological Response of Relapse Subjects That Re-start Treatment With Cyclosporine and/or Eltrombopag
Time Frame: At 1, 2, 3, 6 and 12 months and yearly thereafter
Reporting Status: Not Posted

7. Secondary Outcome: Freedom From h-ATG
Time Frame: At 1, 2, 3, 6 and 12 months and yearly thereafter
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Participants With Severe Aplastic Anemia in Early Initiation of Cyclosporine and Eltrombopag
All-Cause Mortality (participants affected / at risk) | 1/39
Serious Adverse Events (participants affected / at risk) | 24/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Severe Aplastic Anemia in Early Initiation of Cyclosporine and Eltrombopag (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
reversal of ileostomy (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Serum sickness (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (3)
Bone infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Covid-19 infection (Infections and infestations) | 1 (1)
Enterocolitis (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (4)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Increased Intracranial Pressure (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Severe Aplastic Anemia in Early Initiation of Cyclosporine and Eltrombopag (N=39)
Anemia (Blood and lymphatic system disorders) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (17)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chest pressure (right) (Cardiac disorders) | 1 (1)
Chest Tighness (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 11 (16)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (3)
Ear pressure (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Thyroid nodule (Endocrine disorders) | 2 (2)
Anemic Retinopathy (Eye disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Conjunctival Hemorrhage (Eye disorders) | 2 (2)
Diplopia (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Eye Drainage (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eye redness (Eye disorders) | 3 (3)
Flashing lights (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 2 (2)
Inflamed Conjunctiva (Eye disorders) | 2 (2)
Papilledema (Eye disorders) | 1 (1)
Periorbital edema (Eye disorders) | 1 (1)
Pinkish Conjunctiva (Eye disorders) | 2 (2)
Scleral Icterus (Eye disorders) | 1 (1)
Strabismus (Eye disorders) | 1 (1)
Subconjunctival Hemorrhage (Eye disorders) | 2 (2)
Yellow Eyes (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 11 (13)
Acid Reflux (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 3 (3)
Anal pain (Gastrointestinal disorders) | 1 (2)
Bleeding gums (Gastrointestinal disorders) | 8 (13)
Bleeding Lips (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 10 (11)
Dental caries (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 14 (17)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Emesis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (6)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Gum inflammation (Gastrointestinal disorders) | 5 (5)
Gum Swelling (Gastrointestinal disorders) | 4 (4)
Gum tenderness (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 2 (2)
Lip Lesion (Gastrointestinal disorders) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 15 (23)
Oral Blisters (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 3 (3)
Oral pain (Gastrointestinal disorders) | 1 (1)
oropharyngeal bleeding (Gastrointestinal disorders) | 1 (2)
Palate hypertrophy (Gastrointestinal disorders) | 1 (1)
Paracolic fluid (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 4 (4)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Rectal wall thickening (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 5 (5)
Stomatitis (inflamed and sore mouth) (Gastrointestinal disorders) | 1 (1)
Swollen gingival (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (17)
Ankle edema (General disorders) | 1 (1)
Aphthous ulcer (General disorders) | 1 (1)
Chills (General disorders) | 19 (20)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 12 (13)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (9)
Fever (General disorders) | 18 (20)
Flu like symptoms (General disorders) | 1 (1)
generalized achiness (General disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Injection site reaction (General disorders) | 5 (5)
Knee Pain (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 6 (6)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Side Pain (General disorders) | 1 (1)
Thigh pain (General disorders) | 1 (1)
Yellow Eyes (Hepatobiliary disorders) | 4 (5)
Hives (Immune system disorders) | 1 (2)
petechial rash (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (2)
Anorectal infection (Infections and infestations) | 1 (2)
Covid-19 infection (Infections and infestations) | 4 (4)
Folliculitis (Infections and infestations) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
Herpes simplex virus (Infections and infestations) | 1 (1)
Human papillomavirus (Infections and infestations) | 1 (1)
Klebsiella pneumoniae positive (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4)
Skin infection (Infections and infestations) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1)
Tick Bite (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Ankle Injury (Injury, poisoning and procedural complications) | 1 (1)
Bleeding from Skin Biopsy site (Injury, poisoning and procedural complications) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Glass Splinter (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4)
Petechiae (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 22 (43)
Alkaline phosphatase increased (Investigations) | 6 (6)
Anemia (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 18 (28)
Bilirubin, Direct increased (Investigations) | 21 (26)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 28 (44)
Blood lactate dehydrogenase increased (Investigations) | 30 (39)
C-reactive protein increase (Investigations) | 2 (2)
Creatine Kinase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (24)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Haptoglobin decreased (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 12 (12)
Platelet count decreased (Investigations) | 11 (12)
prothrombin time Increased (Investigations) | 1 (1)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 20 (33)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Blood urea nitrogen increase (Metabolism and nutrition disorders) | 2 (2)
Chloride increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperchloremia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 7 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 10 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 25 (38)
Hyponatremia (Metabolism and nutrition disorders) | 10 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Iron overload (Metabolism and nutrition disorders) | 15 (15)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1)
Phosphorus decreased (Metabolism and nutrition disorders) | 1 (1)
Ankle pain (right) (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Elbow Pain (right) (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Growth suppression (Musculoskeletal and connective tissue disorders) | 1 (1)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (20)
Lethargy (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 8 (8)
Seizure (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 4 (4)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Flat Affect (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6)
Jittery (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
sexual dysfunction (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 3 (4)
Hematuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Suprapubic pain (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 2 (2)
Voiding Dysfunction (Renal and urinary disorders) | 1 (1)
Acute Prostatitis (Reproductive system and breast disorders) | 1 (1)
Epididymitis (testicle pain) (Reproductive system and breast disorders) | 1 (1)
Hematochezia (Reproductive system and breast disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (2)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Prostate Calcification (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (13)
Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Jaw Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinovirus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Subglottic Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ashen Pallor (Skin and subcutaneous tissue disorders) | 2 (2)
bilateral hyperpigmented lesions (oral) (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 9 (9)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 3 (3)
Icterus (Skin and subcutaneous tissue disorders) | 2 (2)
Keratotic growth (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritic rash (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Shoulder Nodule (left) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 11 (11)
Yellow Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 20 (21)
Hypotension (Vascular disorders) | 9 (10)
Sinus tachycardia (Vascular disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT04304820/Prot_SAP_000.pdf